CLINICAL TRIAL: NCT00535600
Title: Effects of Bariatric Surgery on Changes in Insulin Secretion and Insulin Action
Brief Title: Effects of Bariatric Surgery on Insulin
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907226; 07-DK-N226
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-03-19

CONDITIONS: Obesity; Bariatric Surgery; Gastric Bypass; Weight Loss; Hyperglycemia
Keywords: Bariatric Surgery; Insulin Action; Insulin Secretion; Insulin Resistance; Gut Hormones; Obesity
MeSH Terms: conditions — Obesity; Weight Loss; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, conducted at the NIH Clinical Research Unit (CRU) at the Phoenix Indian Medical Center, will compare the effects of two methods of bariatric surgery, the adjustable BAND and Roux-en-Y gastric bypass, on insulin. Bariatric surgery is a treatment for achieving and maintaining weight loss. The study will look at how this surgery might improve how insulin (a hormone important for regulating blood sugar levels) is made and works in the body and the possible role of changes in other hormones produced by the gut (stomach and intestines).

People between 18 and 50 years of age who are scheduled to have either laparoscopic adjustable BAND or Roux-en-Y gastric bypass surgery may be eligible for this study. Candidates are screened about 4 to 6 weeks before their surgery with a medical history, blood tests and an oral glucose tolerance test for diabetes.

Participants spend 4 days at the CRU or 2 days overnight and an out-patient visit approximately 4 to 6 weeks before their surgery and again 3 to 6 weeks after their surgery. They return for a 4-6 hour visit at the CRU at 6 months, 1 and 2 years after surgery and for half-day outpatient visits at 3, 4 and 5 years after surgery for the following procedures:

* Blood and urine tests, including a pregnancy test for women. (4-day and 2-day admissions and years, 3, 4 and 5)
* DEXA, an x-ray scan to determine body fat content. (4-day and 2-day admissions and years, 3, 4 and 5)
* MRI scan to measure fat tissue in the abdomen. (4-day and 2-day admissions and years, 3, 4 and 5)
* Intravenous (I.V.) glucose tolerance test for risk of obesity and diabetes. A sugar solution is given through a needle in a vein of one arm and blood samples are drawn through another needle in a vein in the other arm. (4-day admissions)
* Meal test to measure blood sugar and insulin and gut hormone levels after a meal. After an I.V. line is placed in an arm vein, the subject eats breakfast over 20 minutes. Blood samples are collected halfway through the meal, at the end of the meal, and at 15, 30, 60, 90, 120 and 180 minutes after completing the meal. Subjects fill out questionnaires on feelings of hunger and fullness before, during and after the meal test. (4-day and 2-day admissions)
* Glucose clamp test to measure the effect on the body of insulin given through a vein. An I.V line is placed in a vein in the arm and in a vein of the hand on the other side of the body. While insulin is infused through one I.V., blood sugar levels are checked every 5 minutes and a sugar solution is given into a vein as needed. A radioactive sugar is also infused very slowly over 4 hours to determine how much sugar the body produces by itself. (4-day admissions)

DETAILED DESCRIPTION:
Bariatric surgery is a treatment for obesity that, in many cases, also improves fasting blood sugar levels even in patients with type 2 diabetes (T2DM) - within days or weeks after surgery . Both inability to use insulin (insulin resistance) and inability to make enough insulin when needed (impaired insulin secretion) must be present for T2DM to occur, and both have been reported to improve after bariatric surgery. It is generally thought that the immediate improvement in blood sugar levels, including remission of T2DM or "prediabetes" in many patients, following bariatric surgery is due to the markedly reduced intake of calories. However, it is not known why blood sugar levels before and after meals tend to improve earlier and to a greater extent in patients who have a Roux en-Y gastric bypass (RYGB) procedure than in patients who have either the adjustable gastric banding (BAND) or sleeve gastrectomy (SG) procedure. It has been proposed that the surgical alteration of the gut and subsequent re-routing of food that occurs with RYGB procedure results in unique changes in how the gut and pancreas (the organ that secretes insulin) respond to food and that these changes are also related to improved insulin resistance and/or secretion.

The purpose of this protocol is to study, before and after surgery, volunteers who either have normal or impaired ("pre-diabetic") blood sugar regulation and who have been approved to undergo either elective RYGBP, BAND or SG bariatric surgery (n=16 each per surgery group, total = 48 individuals with normal blood sugars; n= 10 each per surgery group, total = 30 individuals with prediabetes). The primary aims are to compare the early effects of the BAND, SG and RYGBP procedures on: a) the ability to maintain blood sugar levels, b) how much insulin is made (secretion) and works (insulin action) in the body, and c) responses of gut and pancreas hormones to a meal test before any significant weight loss occurs after surgery. To achieve these goals, we initially will screen volunteers at the NIH Clinical Research Unit in Phoenix approximately 4-6 weeks prior to surgery (1-day outpatient visit) to determine oral glucose tolerance status (OGTT). Within 3 weeks (1-4 weeks prior to surgery), subjects will then be admitted (4-day in-patient stay) or a 2 day overnight stay and an outpatient (4-6 hour) visit to measure weight, body fatness (DXA scan), waist circumference, insulin resistance, insulin secretion, fasting blood sugar and hemoglobin A1c (HbA1c; a substance that indicates how well the body keeps overall blood sugar levels in a normal range), and plasma hormone responses of the gut and pancreas to a standard meal test. These measurements will be repeated at 3-6 weeks following surgery.

Secondary aims are to: 1) compare long-term effects (up to 5 years) of BAND, SG or RYGBP surgery on fasting blood sugar and HbA1c levels, 2) determine if these levels are related to the responses of gut and pancreas hormones during a meal test, and 3) determine whether pre-op or early post-op measures of insulin secretion, insulin action, or responses of gut and pancreas hormones to a meal can predict long-term levels of fasting blood sugar and HbA1c after accounting for changes in weight or body fat. To achieve these goals, subjects will return to the NIH CRU (out-patient, 4-6 hour visit) at 6, 12, and 24 months after surgery to have repeat measurements of body weight, fatness (DXA, non-contrast MRI of waist and thigh), waist circumference, fasting blood sugar and HbA1c levels and the gut and pancreatic hormone responses to a meal test. Thereafter, subjects will have annual outpatient measurements of body weight, body fat and fasting blood sugar and HbA1c levels at 3, 4 and 5 years after surgery.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must initially qualify for bariatric surgery according to current NIH guidelines, which require the presence of either morbid obesity alone (BMI greater than 40 kg/m(2)) or a BMI greater than 35 kg/m(2) along with at least 2 other co-morbidities.
* Patients with conditions such as sleep apnea, mild steatohepatitis, GERD, asthma (not requiring oral steroids) and osteoarthritis can be considered for participation.
* Subject with undiagnosed diabetes (2-h glucose greater than 200 mg/dl during initial screening OGTT) will be included in the IGR group ONLY IF BOTH fasting plasma glucose is less than 126 mg/dl and HbA1c is less than 7 percent, suggesting early T2DM.
* Subjects must be at least 18 years of age and less than 150 kg body weight.
* Males and females of all ethnic minorities will be included.

EXCLUSION CRITERIA:

Because of the indications for bariatric surgery, many potential subjects will have underlying co-morbidities associated with obesity. For this protocol, subjects will be excluded for the following:

* Current smoking
* Previously diagnosed diabetes
* Other endocrine disorders, such as Cushing's disease, pituitary disorders, and thyroid disease
* Significant hepatic or renal disease (ALT and AST greater than 3-fold above upper limit of normal range, cirrhosis, active hepatitis B or C, serum creatinine greater than 1.5 mg/dl or presence of protein in urine dipstick)
* Active tuberculosis (self-report)
* Major pulmonary disorders including physician diagnosed chronic obstructive pulmonary diseases other than obstructive sleep apnea
* Cardiovascular diseases, including coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
* Hypertension (according to the World Health Organization diagnostic criteria), treated or uncontrolled
* Gastrointestinal disease, including inflammatory bowel diseases (e.g. Crohn's disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active)
* Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis
* Psychiatric conditions or behavior or current alcohol or illicit drug use that would be incompatible with safe and successful participation in this study
* Recent use (within 30 days) of anorexiant medications, antibiotics, contraceptives or fertility drugs or recent use (within 5 days) of anti inflammatory agents
* Pregnancy or breastfeeding (to avoid radiation exposure to fetus or nursing infant)

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-09-21; Study Completion 2014-03-19

CONTACTS AND LOCATIONS:
Overall Officials: Joy C Bunt, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Pontiroli AE, Folli F, Paganelli M, Micheletto G, Pizzocri P, Vedani P, Luisi F, Perego L, Morabito A, Bressani Doldi S. Laparoscopic gastric banding prevents type 2 diabetes and arterial hypertension and induces their remission in morbid obesity: a 4-year case-controlled study. Diabetes Care. 2005 Nov;28(11):2703-9. doi: 10.2337/diacare.28.11.2703. PMID 16249543
- [Background] Ferchak CV, Meneghini LF. Obesity, bariatric surgery and type 2 diabetes--a systematic review. Diabetes Metab Res Rev. 2004 Nov-Dec;20(6):438-45. doi: 10.1002/dmrr.507. PMID 15386803